CLINICAL TRIAL: NCT01781117
Title: Prognostic Value of the Urinary Nerve Growth Factor (NGF) in the Patients With Benign Prostatic Hyperplasia (BPH) Who Undergo Holmium Laser Enucleation of the Prostate (HoLEP)
Brief Title: Prognostic Value of the Urinary Nerve Growth Factor in the Patients With Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KYU-SUNG LEE (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Sponsor-Investigator, KYU-SUNG LEE, Professor, M.D, Ph.D, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-11-013
Record Dates: First submitted 2013-01-21; First posted 2013-01-31 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Benign Prostatic Hypertrophy With Outflow Obstruction; Overactive Detrusor
Keywords: Benign prostatic obstruction (BPO); Detrusor overactivity (DO); Urinary nerve growth factor (NGF)
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HoLEP group (Experimental): Holmium Laser Enucleation of the Prostate (HoLEP)
  Interventions: Procedure: Holmium Laser Enucleation of the Prostate (HoLEP); Device: Holmium laser enucleation system and morcellator

INTERVENTIONS:
Procedure: Holmium Laser Enucleation of the Prostate (HoLEP) — Enucleation of the enlarged nodule of prostate and morcellation of the resected tissue.
Device: Holmium laser enucleation system and morcellator — Holmium laser enucleation and morcellation

SUMMARY:
Persistent detrusor overactivity (DO) after transurethral prostatectomy results in symptomatic failure in more than one third of the patients. Storage symptoms are major complaints in the early postoperative period after Holmium Laser Enucleation of the Prostate (HoLEP). Levels of the urinary nerve growth factor (NGF), produced by bladder urothelium and smooth muscle, are increased in the patients with overactive bladder (OAB), and decreased after the OAB symptoms were improved. Also, urinary NGF levels are increased in patients with benign prostatic obstruction (BPO), but the changes of the NGF levels after relief of the BPO by the medical or surgical treatment have not been fully investigated. If the elevated urinary NGF levels are reduced after successful surgical treatment of BPO, measurement of urinary NGF could be a useful objective tool to assess the therapeutic outcomes of the operation.

The aims of this study are to measure the urinary NGF levels in patients with BPO and to compare the results between the patients with detrusor overactivity (DO) and without detrusor overactivity (Non-DO), average 2 weeks before Holmium Laser Enucleation of the Prostate (HoLEP) procedure. After HoLEP, urinary NGF levels are rechecked at the periods of postoperative 3 months and 6 months, and compare changes between the two groups.

DETAILED DESCRIPTION:
* Investigators are going to enroll age-matched control group and measure the urinary NGF levels as a baseline value (30 males).
* Investigators are going to enroll BPO patients group (DO group 50 and Non-DO group 50 patients).
* Administration of the anti-cholinergic agents was reported to decrease urinary NGF levels. Investigators are going to try to avoid the effect of anti-muscarinic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 50 yrs or greater
* International prostatic symptom score >= 12
* Bladder outlet obstruction confirmed by pressure-flow study (BOOI > 20)
* Ability and willingness to correctly complete the micturition diary and questionnaire
* Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

* Patients with urologic malignancies such as prostate cancer and bladder cancer
* Patients underwent urethral, prostate surgery
* Patients with urethral stricture or bladder diverticulum or bladder neck contracture
* Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2013-02; Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Difference in the baseline urinary NGF level between patients with and without detrusor overactivity at 6 months after HoLEP procedure | 6 months after HoLEP procedure

SECONDARY OUTCOMES:
Difference in the IPSS (International Prostate Symptom Score) and uroflowmetry results between the patients with or without detrusor overactivity | 6 months after HoLEP procedure

OTHER OUTCOMES:
Difference in the serum PSA (Prostate Specific Antigen) level between the patients with or without detrusor overactivity | 6 months after HoLEP procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea